CLINICAL TRIAL: NCT00526396
Title: Multicenter Randomized Phase III Study Comparing Fixed Doses Versus Toxicity Adjusted Dosing of Cisplatin and Etoposide for Patients With Small Cell Lung Cancer.
Brief Title: STAD-1 Small Cell Lung Cancer Toxicity Adjusted Dosing Study
Acronym: STAD-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAD-1; 2006-003995-36 (EudraCT Number)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Small Cell Lung Cancer
Keywords: chemotherapy; toxicity adjusted dose
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): standard fixed doses
  Interventions: Drug: cisplatin; Drug: etoposide
- B (Experimental): toxicity adjusted dosing
  Interventions: Drug: cisplatin; Drug: etoposide

INTERVENTIONS:
Drug: cisplatin — 80 mg/m2 on day 1 for 6 cycles
  Arms: A
Drug: etoposide — 100 mg/m2 on days 1,2,3 for 6 cycles
  Arms: A
Drug: cisplatin — cisplatin on day 1 for 6 cycles, starting dose 80 mg/m2, toxicity adjusted after first cycle
  Arms: B
Drug: etoposide — etoposide on days 1,2,3 for 6 cycles, starting dose 100 mg/m2, toxicity adjusted dosing after first cycle
  Arms: B

SUMMARY:
The purpose of this study is to compare the activity of fixed doses of cisplatin and etoposide with toxicity adjusted dosing of the same drugs in the first-line treatment of small cell lung cancer.

DETAILED DESCRIPTION:
The standard treatment for advanced small cell lung cancer (SCLC) is combination chemotherapy of cisplatin or carboplatin with etoposide. Standard fixed doses of this combination have been based on calculating a patient's body surface area. This method of dose calculation has been shown to be poorly correlated with the activity of many chemotherapy drugs, and some patients do not obtain adequate levels of the drug in their circulation. Recent reports suggest that patients who have a very high tolerability to chemotherapy (without significant toxicity), are at risk for having less effectiveness of the therapy. This study will compare fixed doses of standard chemotherapy with a new strategy of the same chemotherapy with doses that will be adjusted according to the toxicity observed.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic diagnosis of small cell lung cancer
* Extensive disease according to VALG classification
* One or more target lesions.
* Performance status (ECOG) 0 or 1
* Age <70 years.
* Patients with asymptomatic cerebral metastases are eligible
* Patients who have completed treatment with radiation therapy at least 4 weeks prior to enrollment are eligible
* Written informed consent

Exclusion Criteria:

* Previous chemotherapy
* Previous or concomitant malignant neoplasm (excluding adequately treated baso or spinocellular skin carcinoma or carcinoma in situ of the cervix)
* Neutrophil < 2000/mm3, platelets < 100,000/mm3, haemoglobin < 10 g/dl
* Creatinine > 1.5 x the upper normal limits
* GOT and/or GPT > 2.5 and/or Bilirubin > 1.5 times the upper normal limits in absence of hepatic metastases
* GOT and/or GPT > 5 and/or Bilirubin > 3 times the upper normal limits in presence of hepatic metastases
* Any concomitant pathology that would, in the investigator's opinion, contraindicate the use of the drugs in this study
* Hypersensitivity to darbepoetin alpha, to r-HuEPO or their components
* Uncontrolled hypertension.
* Inability to provide informed consent.
* Inability to comply with follow-up

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-09; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
objective response | after 3 and 6 cycles of chemotherapy

SECONDARY OUTCOMES:
toxicity | during and after each treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — S.G. Moscati Hopital, Avellino, Italy, Division of Medical Oncology; Massimo Di Maio, M.D., Principal Investigator — Giannettasio Hospital, Department of Oncology and Hematology; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D, Principal Investigator — Second University of Naples, Italy; Chair of Medical Statistics
Locations (12):
- Italy (12):
  - Azienda Sanitaria S. Giuseppe Moscati, Monteforte Irpino, AV
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Casa di Cura La Maddalena S.p.A., Dipartimento Oncologico, Palermo, PA
  - Istituto Oncologico Veneto, Padua, PD
  - Ospedale E. Morelli, Sondalo, SO
  - Ospedale San Lazzaro, Alba
  - Ospedale Mater Domini, Catanzaro
  - Ospedale L. Sacco Polo Universitario, Milan
  - Istituto Nazionale dei Tumori, Napoli
  - Ospedale Cotugno, Napoli
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Ospedale Maggiore, Trieste

REFERENCES:
- [Derived] Morabito A, Daniele G, Costanzo R, Favaretto AG, Filipazzi V, Rossi A, Gebbia V, Castiglione F, Cavanna L, Maiello E, Sandomenico C, Bonanno L, Piazza E, Maione P, Piccirillo MC, Di Maio M, Rocco G, Gallo C, Perrone F, Gridelli C. A multicenter, randomized, phase 3 trial comparing fixed dose versus toxicity-adjusted dose of cisplatin + etoposide in extensive small-cell lung cancer (SCLC) patients: The Small-cell-lung cancer Toxicity Adjusted Dosing (STAD-1) trial. Lung Cancer. 2017 Jun;108:15-21. doi: 10.1016/j.lungcan.2017.02.016. Epub 2017 Feb 27. PMID 28625627